CLINICAL TRIAL: NCT04639622
Title: GENetic Fronto Temporal Dementia Initiative in Lille
Acronym: GENFI-LILLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018_22; 2018-A02579-46 (Other: ID-RCB)
Record Dates: First submitted 2019-04-26; First posted 2020-11-20 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Frontotemporal Dementia
Keywords: Frontotemporal Dementia; Biomarker; Social cognition; Genetic mutation
MeSH Terms: conditions — Frontotemporal Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- asymptomatic at-risk individual (Other): First-degree relative of a family member affected with the frontotemporal dementia.
  Interventions: Diagnostic Test: Investigation procedures
- symptomatic individual (Other): Patient who has been clinically diagnosed by a neurologist as having frontotemporal dementia or a disorder in the FTD spectrum
  Interventions: Diagnostic Test: Investigation procedures

INTERVENTIONS:
Diagnostic Test: Investigation procedures — All participants will be assessed longitudinally with a set of clinical evaluation, neuropsychiatric and cognitive assessments, imaging (MRI and PET scans) and biosample (CSF, blood samples)

SUMMARY:
GENFI Lille is a French cohort that belongs to the international initiative GENFI2, a five year longitudinal biomarker cohort study of genetic FTD and its associated disorders (including MND/ALS) investigating members of families with a known mutation in GRN or MAPT or an expansion in C9orf72 (including those affected with the disorder as well as at-risk members of families).

DETAILED DESCRIPTION:
The purposes of this study is :

* to improve characterization of symptomatic FTD patients or presymptomatic subjects at risk of genetic FTD
* to develop markers indicative of the optimal time to start disease-modifying therapy, based on the proximity to clinical onset.
* to develop markers of disease progression that can be used as outcome measures.
* to derive sample size estimates for clinical trials.

Participants will include those affected with the disorder as well as at-risk members of families (both mutation carriers and non-carrier first-degree relatives who will serve as a control group).

All participants will be assessed longitudinally with a set of clinical, neuropsychiatric, cognitive, imaging and biosample protocols.

ELIGIBILITY:
Inclusion Criteria:

* The participant must be 18 years old or older.
* The participant must be a member of a family with a known pathogenic mutation in the GRN or MAPT genes, or with a pathogenic expansion in the C9orf72 gene :

  * An affected member is one who has been clinically diagnosed by a neurologist as having frontotemporal dementia or a disorder in the FTD spectrum.
  * An at-risk member is one who is a first-degree relative of a family member affected with the disease.
  * Pathogenicity of a GRN or MAPT mutation is defined by those included within the GENFI list of FTD mutation. If a novel mutation is discovered that is likely to be pathogenic and has not yet been included within the FTD mutation database then the GENFI Genetics Core will decide on inclusion. Please send an email to the GENFI Trials Team at genfi@ucl.ac.uk.
  * A pathogenic C9orf72 expansion is defined as greater than 30 repeats. Intermediate expansions are not considered pathogenic.
  * Participants from one of the small number of families around the world in which 2 (or more) pathogenic mutations have been found should not be included in GENFI.
* If the participant is demented or cognitively impaired there must be an available caregiver that can escort them.
* The participant must have an identified informant.
* The participant must be fluent in the language of their country of assessment.
* The participant accepts that genetic analysis will be carried out on his/her blood samples, and that no results will be available neither for the investigator nor for the participant.

Exclusion Criteria:

* Participant has another medical or psychiatric illness that would interfere in completing assessments.
* Contraindications to FDG-PET (allergy to FDG…)
* Participant is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-23 (Actual); Primary Completion 2025-04-23 (Estimated); Study Completion 2026-04-23 (Estimated)

PRIMARY OUTCOMES:
Difference of the proportion of symptomatic FTD patients or presymptomatic subjects at risk of genetic FTD | each year during 2 years
  Characterization of patients and describe multi characteristics of disease

CONTACTS AND LOCATIONS:
Overall Officials: Thibaud LEBOUVIER, MD, Ph, Principal Investigator — CHU de Lille
Locations (1):
- Hôpital Roger Salengro, CHRU de Lille - CMRR, Lille, France

IPD SHARING:
Plan to Share IPD: No